CLINICAL TRIAL: NCT05232227
Title: Primaquine Double Dose for Radical Cure of Plasmodium Vivax in Colombia
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Trial terminated by funder
Sponsor: University of California, San Francisco (Other)
Collaborators: Pan American Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-34422
Record Dates: First submitted 2021-11-18; First posted 2022-02-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Malaria, Vivax; Relapse
Keywords: Plasmodium vivax; Radical cure regimen; Primaquine double dose (PQdd); Colombia
MeSH Terms: conditions — Malaria, Vivax; Recurrence | interventions — Primaquine

STUDY DESIGN:
Masking Description: A randomized open-label superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard regimen Primaquine single dose over 14 days (Active Comparator): The standard regimen consists of administering Chloquine Phosphate 10 mg/kg on days 1 and 2, and 5 mg/kg on day 3 plus Primaquine Phosphate 3.5 mg/kg divided over 14 days (0.25mg/kg/day)
  Interventions: Drug: Primaquine single dose over 14 days
- Treatment regimen Primaquine double dose over 14 days (Experimental): The treatment regimen consists of administering Chloquine Phosphate 10 mg/kg on days 1 and 2, and 5 mg/kg on day 3 plus Primaquine Phosphate 7 mg/kg divided over 14 days
  Interventions: Drug: Primaquine double dose over 14 days

INTERVENTIONS:
Drug: Primaquine double dose over 14 days — Primaquine Phosphate tablets New Drug Application (NDA): 008316 Company: SANOFI AVENTIS US Chloroquine Phosphate tablets
  Other Names: Primaquine Phosphate tablets
  Arms: Treatment regimen Primaquine double dose over 14 days
Drug: Primaquine single dose over 14 days — Primaquine Phosphate tablets New Drug Application (NDA): 008316 Company: SANOFI AVENTIS US
  Other Names: Primaquine Phosphate tablets
  Arms: Standard regimen Primaquine single dose over 14 days

SUMMARY:
Primaquine (PQ) is the only widely available treatment to prevent P. vivax relapses. World Health Organization recommends increased PQ doses in East Asia and Oceania, frequently relapsing strains. In 2005, the Centers for Diseases Control and Prevention began also recommending higher dose PQ to treat infections from all parts of the world.

In Latin America, PQ for a radical cure has been largely implemented as 3.5 mg/kg over 14 days (standard dose, long-course, PQsd14) or 3.5 mg/kg over 7 days (short-course, or PQsd7) in combination with chloroquine (CQ). A recent randomized controlled trial in Brazil showed that a 7 mg/kg double dose regimen over 14 days (PQdd14) was superior in preventing relapses compared to the standard of care regimen in Brazil of 3.5 mg/kg over 7 PQsd7 Direct Observed Therapy (DOT) and PQsd7 without DOT and with or 14 days PQsd14 with DOT (92% versus 66% were relapse-free in the 6-month follow-up in adjusted analyses). These data were presented at the 2019 PAHO Malaria Technical Advisory Group (TAG) meeting. To inform whether there should be a policy change by Panamerican Health Organization, the Malaria TAG recommended more evidence from the results of another trial to confirm the efficacy of high versus low-dose PQ. This project aims to generate the necessary evidence to inform a policy decision regarding high-dose PQ.

Impact Malaria (IM) proposes to conduct another trial, per the PAHO Malaria TAG's recommendation, assessing the efficacy of high-dose PQ compared to low-dose PQ. The objective is to compare a standard regimen, which in Colombia is PQsd14 (3,5mg/kg divided in 14 days), to a double dose alternative PQ 7 mg/kg double dose regimen over 14 days (PQdd14).

DETAILED DESCRIPTION:
Malaria due to Plasmodium vivax (P. vivax) is still a public health challenge in the Americas. In recent years, the rate of decline in the incidence of P. vivax malaria has stalled in the Americas. To address this challenge and support countries in Latin America & the Caribbean (LAC) aiming for malaria elimination, effective treatment strategies against P. vivax are needed. Primaquine (PQ) is the only widely available treatment to prevent P. vivax relapses. WHO recommends increased PQ doses in East Asia and Oceania, where strains are frequently-relapsing. In 2005, the Centers for Diseases Control and Prevention (CDC) began also recommending higher dose PQ to treat infections from all parts of the world.

In Latin America, PQ for a radical cure has been largely implemented as 3.5 mg/kg over 14 days (standard dose, long-course, PQsd14) or 3.5 mg/kg over 7 days (short-course, or PQsd7) in combination with chloroquine (CQ). A recent randomized controlled trial in Brazil showed that a 7 mg/kg double dose regimen over 14 days (PQdd14) was superior in preventing relapses compared to the standard of care regimen in Brazil of 3.5 mg/kg over 7 PQsd7 Direct Observed Therapy (DOT) and PQsd7 without DOT and with or 14 days PQsd14 with DOT (92% versus 66% were relapse-free in the 6-month follow-up in adjusted analyses). These data were presented at the 2019 PAHO Malaria Technical Advisory Group (TAG) meeting.

To inform whether there should be a policy change by PAHO, the Malaria TAG recommended more evidence from the results of another trial to confirm the efficacy of high versus low-dose PQ. This project aims to generate the necessary evidence to inform a policy decision regarding high-dose PQ.

Impact Malaria (IM) proposes to conduct another trial, per the PAHO Malaria TAG's recommendation, assessing the efficacy of high-dose PQ compared to low-dose PQ. The objective is to compare a standard regimen, which in Colombia is PQsd14 (3,5mg/kg divided in 14 days), to a double dose alternative: PQ 7 mg/kg double dose regimen over 14 days (PQdd14).

PQ, the mainstay for a radical cure for P. vivax, induces a dose-dependent acute hemolytic anemia in individuals with Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency. Where available, WHO recommends G6PD deficiency testing prior to PQ administration. In LAC countries, where G6PD deficiency testing is not widely available, Low-dose PQ without G6PD deficiency testing has been a standard approach regimen for more than 60 years. Low prevalence of G6PD deficiency, a predominance of less severe variants, and the absence of historical reports of hemolysis with the 14-day Low-dose regimen have allowed for this unsystematic, standard approach without testing. Nevertheless, PAHO promotes pharmacovigilance and early recognition of signs of hemolysis to enable stopping PQ to prevent more severe outcomes. However, countries are not implementing these approaches systematically. Improved pharmacovigilance and G6PD deficiency testing may be needed if higher dose PQ regimens are recommended, as these regimens have a higher potential to cause severe hemolysis and other adverse events. Higher dose regimens may also be less well tolerated, and therefore compromise adherence. At the same time, where quality G6PD deficiency testing is not reliable or available, a risk-benefit assessment may suggest that the benefits of using high dose PQ without G6PD deficiency testing may still outweigh such risks.

Following current recommendations that G6PD deficiency testing is conducted prior to PQ or TQ administration, low G6PD activity, measured by a quantitative rapid test (Standard Diagnostics (SD) Biosensor), will be an exclusion criterion. As the primary goal of this study is to assess the efficacy of the new regimens, all regimens will be administered by directly observed therapy (DOT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥5 years
* Fever (T≥37.5 ⁰C, oral) and/or history of fever in the previous 48 hours
* P. vivax mono-infection
* Normal G6PD status using Biosensor™ (SD Bioline, ROK) (G6PD activity ≥ 70% of the adjusted male median (AMM))
* Written informed consent
* Living in the study area and willing to be followed for six months

Exclusion Criteria:

* Malaria treatment in the previous 30 days,
* Self-reported chronic disease (including severe cardiac, hepatic, or renal disorders, malnutrition, or HIV),
* Clinically significant concurrent illness,
* Use of medications known to interfere with the pharmacokinetics of PQ or CQ,
* Known hypersensitivity to any of the study drugs,
* Use of an investigational drug within the previous 30 days or five half-lives (whichever was longer),
* History of moderate or severe adverse reaction to any of the study drugs,
* Hemoglobin < 7 g/dL,
* Pregnancy (by urine pregnancy test) or breastfeeding,
* Not able to take oral treatment,
* Signs of severe malaria:

  * Unable to drink
  * Vomiting (more than twice in the previous 24 hours)
  * Recent history of convulsions (one or more in the previous 24 hours)
  * Impaired consciousness
  * Unable to sit or stand
  * Cerebral malaria (unarousable coma)
  * Severe anemia (hematocrit <15% or clinical signs) hemoglobin <5 mg/ml) (Note: we will use hemoglobin less than 7 mg/ml as exclusion criteria)
  * Renal failure (serum creatinine >3 mg/dL or clinical signs)
  * Pulmonary edema
  * Hypoglycemia (blood glucose <40mg/dL or clinical signs)
  * Shock (systolic blood pressure <70 mm Hg in adults; 50 mm Hg in children)
  * Spontaneous bleeding/disseminated intravascular coagulation.
  * Repeated generalized convulsions
  * Acidemia/acidosis (clinical signs)
  * Macroscopic hemoglobinuria
  * Jaundice●

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2023-06-05 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence risk of microscopy-detectable P. vivax infections | 6-month follow-up
  The incidence risk (time to first event) of microscopy-detectable P. vivax infection (sexual and asexual parasitemias), comparing PQdd14 to PQsd14.

SECONDARY OUTCOMES:
relapse efficacy | 6-month follow-up
  The incidence risk of symptomatic, microscopy-detectable P. vivax infection, The incidence risk of severe anemia (Hb < 7g/dl) and/or requiring blood transfusion comparing PQdd14 to PQsd14.
  * The incidence rate (events per person-time) of microscopy-detectable P. vivax infection, comparing PQdd14 to PQsd14.
  * The incidence rate (events per person-time) of symptomatic, microscopy-detectable P. vivax infection, comparing PQdd14 to PQsd14.

IPD SHARING:
Plan to Share IPD: No